CLINICAL TRIAL: NCT01092572
Title: The Effect of Simvastatin on Systemic Inflammation in Adult Cystic Fibrosis Subjects: A Pilot Study
Brief Title: Statins To Treat Adult Cystic Fibrosis
Acronym: CFStatin
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF-Man-Statin-1
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Cystic Fibrosis; Systemic Inflammation
Keywords: cystic fibrosis; adult cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin 40 mg/d (Experimental): simvastatin 40 mg per day taken orally
  Interventions: Drug: Simvastatin
- Sugar pill (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Simvastatin — simvastatin 40 mg per day orally for 12 weeks.
  Arms: Simvastatin 40 mg/d
Drug: placebo — placebo 1 tablet once daily for 12 weeks
  Arms: Sugar pill

SUMMARY:
Cystic fibrosis (CF) is a lethal genetic condition that affects 30,000 children and adults in the United States. Although CF management has improved substantially over the past two decades, there is still no cure and most patients with CF die before reaching their 50th birthday, largely due to lung failure. There is growing evidence that excess lung and blood inflammation that occurs in response to infections in the lungs cause CF patients to be sicker. Simvastatin is a drug that is used to lower cholesterol, but many researchers have found that this drug may also treat blood and lung inflammation. In this study, we will determine whether or not simvastatin can treat blood and lung inflammation in patients with CF and most importantly determine whether or not it can make these patients feel better and have better lung function.

DETAILED DESCRIPTION:
Study Objectives

1. To determine the effect of 12 weeks of 40 mg once daily simvastatin on general inflammatory molecules, IL-6 and CRP in the blood of CF patients.
2. To determine the effect of simvastatin on LPS-related pathway molecules in the blood.
3. To determine the effect of simvastatin on inflammatory pneumo-proteins in the blood.
4. To determine exacerbation and safety data on statins in preparation for a large phase III trial of statins in CF.

Study Endpoints

The primary endpoint will be the quantitative changes in serum levels of CRP.

Secondary endpoints will include:

1. blood biomarkers IL6, LPS related proteins, LPS, LBP, sCD14 and EndoCAb, and pneumoproteins, SPD and CCL18; and molecules such as TNF-α and IL-1beta;
2. changes in FEV1 over 12 weeks ; and
3. exacerbations over 12 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Patients of provincial legal age of majority in British Columbia (≥19 years of age);
2. Confirmed diagnosis of CF based on the following criteria:

   1. One or more clinical features consistent with the CF phenotype
   2. A genotype with identifiable classes I or II CFTR mutations
3. Ability to provide informed consent.
4. Clinically stable at enrollment as assessed by the treating physician.
5. Ability to comply with medication use, study visits and study procedures, such as spirometry, and venipunctures.

Exclusion Criteria:

1. Allergy or clinical reaction to simvastatin.
2. The following abnormal lab values within the last six months or at screening:

   AST/ALT > 1.5 ULN, CK > 1.5 ULN, and eGFR < 40ml/min/1.73m2.
3. Use of intravenous antibiotics or oral quinolones within 14 days of screening.
4. With the exception of Azithromycin the use of oral antibiotics including prophylactic antibiotics (e.g., augmentin, tetracycline, cloxacillin, cephalosporins, trimethoprim/sulfamethoxazole) within 14 days of screening.
5. Initiation of high dose ibuprofen, dornase alpha, hypertonic saline or aerosolized antibiotics within 30 days of screening.
6. On medications that are known to have potential serious interactions with simvastatin (as listed on page 10 of this protocol).
7. Use of systemic corticosteroids within 30 days of screening.
8. Investigational drug use within 30 days of screening.
9. Other major organ dysfunction excluding pancreatic dysfunction.
10. History of lung transplantation or currently on lung transplant list.
11. Pregnant, breast feeding, or if post-menarche female, unwilling to practice birth control during participation in the study.
12. Chronic users of niacin, azole antifungals (itraconazole, ketoconazole, voriconazole), telithromycin, fibric acid derivatives, HIV protease inhibitors, amiodarone, digoxin and/or cyclosporine (to decrease the risk of statin-related myotoxicity).
13. Patients who are colonized or infected with Burkholderia cepacia complex are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | 12 weeks
  The difference in the change in plasma C-reactive protein concentrations from baseline to 12 weeks of treatment between those randomized to simvastatin 40 mg/d and those randomized to placebo

SECONDARY OUTCOMES:
Changes in forced expiratory volume in one second (FEV1) | 12 weeks
  The differences in the above parameters over 12 weeks between those assigned to simvastatin 40 mg/d and those assigned to placebo.
Changes in exacerbation rates | 12 weeks
  The differences in the above parameters over 12 weeks between those assigned to simvastatin 40 mg/d and those assigned to placebo.
Changes in blood pro-inflammatory markers such as IL-6, TNF, IL-1beta, LPS, LBP, sCD14, EndoCAB, SP-D, CCL-18) | 12 weeks
  The differences in the above parameters over 12 weeks between those assigned to simvastatin 40 mg/d and those assigned to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Man, MD, Principal Investigator — University of British Columbia